CLINICAL TRIAL: NCT00333112
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multicenter Safety and Efficacy, Phase 4 Study of VESIcare® (Solifenacin Succinate) or Placebo in Combination With Tamsulosin HCl for the Treatment of Residual OAB Symptoms of Urgency and Frequency in Men VICTOR: VESIcare® In Combination With Tamsulosin in OAB Residual Symptoms
Brief Title: A Study to Evaluate Solifenacin Succinate in Combination With Tamsulosin for the Treatment of Residual Overactive Bladder Symptoms (OAB) in Men.
Acronym: VICTOR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 905-UC-008
Record Dates: First submitted 2006-06-01; First posted 2006-06-02 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Urinary Incontinence
Keywords: Treatment Outcome; Urology; Solifenacin succinate; Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence | interventions — Solifenacin Succinate; Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: solifenacin succinate; Drug: tamsulosin
- 2 (Placebo Comparator)
  Interventions: Drug: tamsulosin; Drug: placebo

INTERVENTIONS:
Drug: solifenacin succinate — Oral
  Other Names: Vesicare®; YM905
  Arms: 1
Drug: tamsulosin — oral
Drug: placebo — oral
  Arms: 2

SUMMARY:
A study to evaluate solifenacin succinate in combination with tamsulosin for the treatment of residual OAB symptoms in men.

DETAILED DESCRIPTION:
A 2 arm study ( 1 Active, 1 Placebo) to evaluate solifenacin succinate in combination with tamsulosin for the treatment of residual OAB symptoms in men

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of Overactive Bladder (OAB)

Exclusion Criteria:

* Current use of antimuscarinic therapy
* Evidence of a urinary tract infection

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2006-05; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Change in micturitions per 24 hours from baseline to end of treatment | 18 weeks

SECONDARY OUTCOMES:
Change in urgency episodes per 24 hours from baseline to end of treatment | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Astellas US Medical Information, Study Director — Astellas Pharma US, Inc.
Locations (70):
- United States (70):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Tuscon, Arizona
  - Atherton, California
  - Beverly Hills, California
  - Buena, California
  - Buena Park, California
  - Carmichael, California
  - Culver City, California
  - Fresno, California
  - Mission Hills, California
  - Modesto, California
  - Orange, California
  - San Bernardino, California
  - San Diego, California
  - Torrance, California
  - Aurora, Colorado
  - Denver, Colorado
  - Wheat Ridge, Colorado
  - Danbury, Connecticut
  - Clearwater, Florida
  - Daytona Beach, Florida
  - Fort Myers, Florida
  - New Port Richey, Florida
  - Orlando, Florida
  - Pembroke Pines, Florida
  - Tallahassee, Florida
  - Wellington, Florida
  - Atlanta, Georgia
  - Blue Ridge, Georgia
  - Marietta, Georgia
  - Roswell, Georgia
  - Sandy Springs, Georgia
  - Snellville, Georgia
  - Coeur d'Alene, Idaho
  - Evansville, Indiana
  - Wichita, Kansas
  - Shreveport, Louisiana
  - Boston, Massachusetts
  - Watertown, Massachusetts
  - Grand Rapids, Michigan
  - Jackson, Mississippi
  - West Orange, New Jersey
  - Endwell, New York
  - Garden City, New York
  - New York, New York
  - Orchard Park, New York
  - Poughkeepsie, New York
  - Rochester, New York
  - Concord, North Carolina
  - Hickory, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Bethany, Oklahoma
  - Norman, Oklahoma
  - Springfield, Oregon
  - Bala-Cynwyd, Pennsylvania
  - Bensalem, Pennsylvania
  - Camp Hill, Pennsylvania
  - Lancaster, Pennsylvania
  - Uniontown, Pennsylvania
  - Mt. Pleasant, South Carolina
  - Simpsonville, South Carolina
  - Nashville, Tennessee
  - Houston, Texas
  - Ogden, Utah
  - Salt Lake City, Utah
  - Virginia Beach, Virginia
  - Mountain Lake Terrace, Washington
  - Spokane, Washington

REFERENCES:
- [Background] Kaplan SA, McCammon K, Fincher R, Fakhoury A, He W. Safety and tolerability of solifenacin add-on therapy to alpha-blocker treated men with residual urgency and frequency. J Urol. 2009 Dec;182(6):2825-30. doi: 10.1016/j.juro.2009.08.023. Epub 2009 Oct 17. PMID 19837435